CLINICAL TRIAL: NCT05372536
Title: Parent-Administered Low-Dose Cytarabine to Children and Adolescents With Cancer at Home - a Feasibility Study
Brief Title: Home Chemotherapy Intervention for Children With Cancer - a Feasibility Study
Acronym: INTACTatHome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Louise Ingerslev Roug, Principal Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LROU0001-1
Record Dates: First submitted 2022-04-25; First posted 2022-05-12 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Supportive Care; Childhood Cancer
Keywords: Home chemotherapy
MeSH Terms: conditions — Neoplasms | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- parent-led home-administered low-dose Cytarabine (Experimental): Parents to the included participants are offered to administer the protocolized low-dose bolus (injection) Cytarabine in their children's CVCs at home. The administration procedure is developed as a simple and safe non-touch technique. The parents receive a video and paper-based guideline and information material followed by a 3-step nurse-led education program. The parents can administer the Cytarabine at home when they (and the child/adolescent) feel safe and comfortable managing the procedure and when the nurses are sure that the parents can manage the procedure at home. The first dose of Cytarabine is always administered at the hospital.
  Interventions: Other: parent-led home-administered low-dose Cytarabine

INTERVENTIONS:
Other: parent-led home-administered low-dose Cytarabine — Parents to the included participants are offered to administer the protocolized low-dose bolus (injection) Cytarabine in their children's CVCs at home. The administration procedure is developed as a simple and safe non-touch technique. The parents receive a video and paper-based guideline and information material followed by a 3-step nurse-led education program. The parents can administer the Cytarabine at home when they (and the child/adolescent) feel safe and comfortable managing the procedure and when the nurses are sure that the parents can manage the procedure at home. The first dose of Cytarabine is always administered at the hospital.

SUMMARY:
Children with cancer undergo intensive treatment with many serious side effects and frequent in- and outpatient visits. Studies show that the frequent hospitalizations are very disruptive to children and their families, who strive to maintain a normal everyday life. The aim of the study is to test a parent-led home-administered low-dose cytarabine intervention that will not compromise the quality of treatment and care, increase the caregiver burden or the experienced symptoms of the children. The methodical approach is based on The Medical Research Council's framework to develop and evaluate complex interventions in health care using both clinical observational methods, participatory methods, surveys and qualitative ethnographic methods. The overall goal of the project is to support and ease the everyday lives of children with cancer and their families during the intensive treatment periods.

DETAILED DESCRIPTION:
This single-arm feasibility study is conducted at Copenhagen University Hospital, Rigshospitalet, in Denmark at the Department of Pediatric Oncology and Hematology.The PI started to recruit participants March 2022. Patients with Acute Lymphoblastic Leukemia (ALL), Philadelphia positive Acute Lymphoblastic Leukemia (PH+ALL) and Lymphoblastic Lymphoma (LBL) are eligible for inclusion if their parents speak and understand Danish or English, able to manage basic treatment and care such as oral medication, mobilization, nutrition, central venous catheter care and practice good personal hygiene. The parents' competences are assessed by the PI in collaboration with a team of project- and ward nurses who know them. Participants are recruited between day 15 and 29 from diagnosis. Parents to eligible participants and adolescents aged 15+ receive oral and written information and provide written informed consent before inclusion. Children and adolescents less than 15 years of age receive oral information and provide oral consent if possible according to their age. Parents to the included participants are offered to administer the protocolized low-dose bolus (injection) Cytarabine in their children's CVCs at home. The administration procedure is developed as a simple and safe non-touch technique. The parents receive a video and paper-based guideline and information material followed by a 3-step nurse-led education program. The parents can administer the Cytarabine at home when they (and the child/adolescent) feel safe and comfortable managing the procedure and when the nurses are sure that the parents can manage the procedure at home. The first dose of Cytarabine is always administered at the hospital.

ELIGIBILITY:
Inclusion Criteria:

- Children/adolescents diagnosed with ALL, LBL or PH+ ALL

Exclusion Criteria:

* If their parents did not understand, read and speak Danish
* If the parents did not manage the children/adolescents' basic care and treatment needs (CVC care, oral medication, hygiene, nutrition, mobilization, ect.)

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | From day 15 (from protocol start) until the last day with low dose cytarabine treatment which depends on protocol stratification and randomization (mean intervention period = 22 weeks)
  Number of families who consent to participate in the study
Attrition rate | From time of obtained consent until end of intervention period (mean intervention period = 22 weeks)
  Number of drop-outs during the intervention
Demand (dose) | From day 38 up to day 167 from protocol start. Four to eight timepoints depending on number of protocolized cytarabine doses (mean intervention period = 22 weeks)
  Number of parent-led home-administered low-dose Cytarabine (total and average)
Education time | From time of obtained consent until start of intervention (2-4 weeks)
  Time (minutes) nurses spent on education for parents before the intervention
Adverse events | From recruitment start to end of intervention (mean intervention period = 22 weeks)
  Severe and non-severe events
Respons rate | Everyday during each four-day-long chemo-cycle to five days after (one to eight cycles are given depending on the specific protocol).The typical intervention period is 22 weeks
  Number of responses on PENAT questionnaire
Respons rate | At the end of each chemo-cycle (day 4, each chemo-cycle is four days). The typical intervention period is 22 weeks
  Number of responses on CMCC and SS questionnaires

SECONDARY OUTCOMES:
Nausea and Vomiting during low-dose Cytarabine treatment (tentative) | Starting day one of the Cytarabine cycle and stops five days after (9 days). Each Cytarabine cycle is four days. There can be from four to eight cycles of Cytarabine in the Protocol.
  Questionnaire (PENAT - measuring chemotherapy induced nausea and vomiting))
Caregiver Demands (tentative) | Day four (and the last day) of each cycle of Cytarabine (each cycle is four days)
  Questionnaire (CMCC: Care of My Child with Cancer)
Satisfaction and safety (tentative) | Day four (and the last day) of each cycle of Cytarabine (each cycle is four days)
  Questionnaire measuring parents and children/adolescents' experience of satisfaction and safety managing the home-administration of Cytarabine)
The family's experience of the intervention of home-administered Cytarabine | Interviews are conducted after end intervention (approximately day 167 since protocol start)
  qualitative interviews with parents and children/adolescents
Adaption, Integration, implementation | Fieldnotes are collected at various timepoints during the in total study/intervention period = 43 weeks
  Qualitative process evaluation of the feasibility areas: Adaption, integration and implementation

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Madsen, Chief nurse, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Louise Ingerslev Roug, Copenhagen, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roug LI, Topperzer MK, Michelsen RT, Jarden M, Wahlberg A, Hjalgrim LL, Hansson H. Development of an intravenous chemotherapy intervention for children and adolescents with cancer administered by their parents at home (INTACTatHome). BMC Health Serv Res. 2023 Jun 20;23(1):664. doi: 10.1186/s12913-023-09613-2. PMID 37340397